CLINICAL TRIAL: NCT00387699
Title: Phase II Trial of Bevacizumab in Combination With Cisplatin/Etoposide and Twice Daily Radiation for Patients With Limited-Stage Small Cell Lung Cancer
Brief Title: Bevacizumab, Cisplatin, Etoposide, and Radiation Therapy in Treating Patients With Limited-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Robert L. Comis, ECOG Group Chair's Office
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000508653; ECOG-E1506
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2008-10

CONDITIONS: Lung Cancer
Keywords: limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Bevacizumab; Cisplatin; Etoposide; Radiotherapy

INTERVENTIONS:
Biological: bevacizumab
Drug: cisplatin
Drug: etoposide
Radiation: radiation therapy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some find tumor cells and help kill them or carry tumor-killing substances to them. Others interfere with the ability of tumor cells to grow and spread. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Drugs used in chemotherapy, such as cisplatin and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving bevacizumab together with cisplatin, etoposide, and radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving bevacizumab together with cisplatin, etoposide, and radiation therapy works in treating patients with limited-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 1-year progression-free survival of patients with limited-stage small cell lung cancer treated with bevacizumab, cisplatin, etoposide, and radiotherapy.

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine the response rate in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive cisplatin IV over 30-60 minutes and bevacizumab IV over 30-90 minutes on day 1 and etoposide IV over 60 minutes on days 1-3. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. During course 1, patients also undergo thoracic radiotherapy twice daily on days 1-5, 8-12, and 15-19.

Patients achieving a complete or partial response or stable disease after the first 4 courses of chemotherapy continue to receive bevacizumab IV over 30-90 minutes on day 1. Treatment with bevacizumab repeats every 21 days for up to 1 year in the absence of disease progression or unacceptable toxicity.

Within 4-6 weeks after blood counts recover from the first 4 courses of chemotherapy, patients achieving a complete or partial response also undergo prophylactic cranial irradiation (PCI) in 10 fractions over 3 weeks.*

NOTE: *Bevacizumab should not be given for 3 weeks prior to or during PCI, but resumed 1 week after completion of PCI.

After completion of study treatment, patients are followed periodically for 10 years.

PROJECTED ACCRUAL: A total of 79 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed small cell lung cancer (SCLC)

  * Limited-stage disease, defined as SCLC confined to ≥ 1 of the following:

    * One hemithorax
    * Ipsilateral supraclavicular fossa
* Measurable disease
* No malignant pleural effusion, contralateral hilar disease, or contralateral supraclavicular disease

  * Minimal pleural effusion visible on CT scan of the chest, but not evident on chest x-ray, allowed
* No completely surgically resected disease
* No CNS disease, including primary brain tumor or brain metastasis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 mg/dL
* Creatinine ≤ 1.5 mg/dL
* Urine protein:creatinine ratio ≤ 0.5 OR 24-hour urine protein < 1,000 mg
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study treatment
* INR ≤ 1.5 (unless on full-dose anticoagulants)
* No active serious infection
* No serious or nonhealing wound
* No ulcer or bone fracture
* No evidence of bleeding diatheses or coagulopathy
* No hemoptysis
* No known hypersensitivity to Chinese hamster ovary cell products and/or other recombinant human antibodies
* No clinically significant cardiovascular disease, including any of the following:

  * Uncontrolled hypertension
  * New York Heart Association class II-IV congestive heart failure
  * Serious cardiac arrhythmia requiring medication
  * Unstable angina pectoris
  * Symptomatic peripheral vascular disease
  * Cerebrovascular accident within the past 6 months
  * Symptomatic heart disease within the past 6 months
  * Myocardial infarction within the past 6 months
  * Unstable angina within the past 6 months
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 4 weeks
* No significant traumatic injury within the past 4 weeks

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior major surgery or open biopsy
* At least 1 week since prior core biopsy
* No prior chemotherapy or radiotherapy for small cell lung cancer
* No concurrent major surgery
* No concurrent palliative local radiotherapy
* No concurrent intensity-modulated radiotherapy
* Concurrent full-dose anticoagulants (e.g., warfarin) allowed provided all of the following criteria are met:

  * INR ≤ 3
  * In-range INR (2-3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin
  * No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2006-10; Primary Completion 2007-10 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Progression-free survival at 1 year

SECONDARY OUTCOMES:
Response rate
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Dowlati, MD, Study Chair — Case Comprehensive Cancer Center; James A. Bonner, MD — University of Alabama at Birmingham